CLINICAL TRIAL: NCT05560217
Title: a Study That Collection of Peripheral Blood Mononuclear Cells From Healthy Subjects
Brief Title: Collection of Peripheral Blood Mononuclear Cells From Healthy Subjects
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2022-115-02
Record Dates: First submitted 2022-09-26; First posted 2022-09-29 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Disease of the Blood
MeSH Terms: conditions — Hematologic Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In accordance with the selection criteria, component blood collection will be carried out and peripheral blood mononuclear cells will be isolated, cryopreserved and in vitro culture of peripheral blood mononuclear cells. Cultivating cells under normal culture conditions or potential drug molecule treatment, observing and recording key parameters such as cell viability, proliferation, apoptosis and functional gene expression, will also provide an important reference for the production of CAR-T cell drugs.

DETAILED DESCRIPTION:
aged 18-40, regardless of nationalities, and had no adverse reactions in blood donation; Weight: male≥50kg, female≥45kg, and 18.5kg/m2≤BMI≤30kg/m2 (BMI =weight（kg）÷height（m）2)；

Blood pressure:

12.0Kpa（90mmHg）≤systolic pressure<18.7Kpa（140mmHg） 8.0Kpa（60mmHg）≤diastolic pressure<12.0Kpa（90mmHg）； Pulse rate: 60 beats/ min ~ 100 beats/ min, the athlete with high-level stamina≥50 beats/ min, normal and tidy rhythm.

Body temperature:36.3-37.2℃; Generally in good condition: no impairment of major organs, including heart, lung, liver, and kidney, no serious or uncontrolled infections, and no history of severe mental illness;

The clinical lab tests must meet the following standards:

Blood routine, blood biochemistry, normal or abnormal liver and kidney function have no clinical significance; Normal testing of coagulation function; Negative for antibody to Hepatitis A Virus (HAV-IgM); Negative for Hepatitis B Virus Surface Antigen (HBsAg); Negative for antibody to Hepatitis C Virus (HCV); Negative for antibody to Human Immunodeficiency Virus (HIV-1 and HIV-2); Negative for Syphilis; Negative for DNA to Epstein-Barr Virus (EBV). Negative for DNA to cytomegalovirus (CMV) . Negative for DNA to B19. Negative for Human T Lymphocytic leukemia Virus (HTLV).

ELIGIBILITY:
Inclusion Criteria:

* aged 18-40, regardless of nationalities, and had no adverse reactions in blood donation;
* Weight: male≥50kg, female≥45kg, and 18.5kg/m2≤BMI≤30kg/m2 (BMI =weight（kg）÷height（m）2)；
* Blood pressure:

12.0Kpa（90mmHg）≤systolic pressure<18.7Kpa（140mmHg） 8.0Kpa（60mmHg）≤diastolic pressure<12.0Kpa（90mmHg）； Pulse rate: 60 beats/ min ~ 100 beats/ min, the athlete with high-level stamina≥50 beats/ min, normal and tidy rhythm.

* Body temperature:36.3-37.2℃;
* Generally in good condition: no impairment of major organs, including heart, lung, liver, and kidney, no serious or uncontrolled infections, and no history of severe mental illness;
* The clinical lab tests must meet the following standards:

Blood routine, blood biochemistry, normal or abnormal liver and kidney function have no clinical significance; Normal testing of coagulation function; Negative for antibody to Hepatitis A Virus (HAV-IgM); Negative for Hepatitis B Virus Surface Antigen (HBsAg); Negative for antibody to Hepatitis C Virus (HCV); Negative for antibody to Human Immunodeficiency Virus (HIV-1 and HIV-2); Negative for Syphilis; Negative for DNA to Epstein-Barr Virus (EBV). Negative for DNA to cytomegalovirus (CMV) . Negative for DNA to B19. Negative for Human T Lymphocytic leukemia Virus (HTLV).

Exclusion Criteria:

* You have diseases in respiratory, circulatory, digestive, urinary, blood, immune, endocrine system or metabolic disorders;
* You have neurological diseases, mental diseases, Creutzfeldt-Jakob disease and have a family medical history or those who have received treatment with tissues or tissue derivatives that may be infected by Creutzfeldt-Jakob pathogen;
* You have chronic skin diseases, especially infectious, allergic or inflammatory systemic skin diseases;
* You have allergic diseases or frequent relapse;
* You have/had malignant tumors or benign tumors cause health problems;
* You have an infectious disease, a carrier of an infectious disease, a suspected infectious disease;
* You have allogeneic tissue organ graft recipients.
* You have undergone the removal of important internal organs such as the stomach, kidneys, spleen, lungs and so on;
* Those who have caused the recipient to have infectious diseases related to blood transfusion.
* You have had minor surgery within 3 months, including appendectomy, eye surgery, etc.; major surgery within 1 year, such as: surgical treatment of gynecological benign tumor, superficial benign tumor, etc.;
* Women in pregnancy or had a miscarriage within 6 months, or post partum and in lactation within 1 year;
* Recovered from Upper respiratory tract infection no longer than one week, or from pneumonia no longer than three months;
* Recovered from Acute pyelonephritis no longer than 3 months, or within the attack period of the urinary tract stones;
* Injuries caused by or wounds contaminated by devices/apparatuses contaminated by blood or tissue fluid or tattooed within one year;
* You have received whole blood and blood component transfusion within 1 year;
* You have got the last vaccination of live attenuated vaccines within 2 weeks including measles, parotitis, or infantile paralysis, or got the last vaccination of live attenuated vaccines within 4 weeks including Rubella Vaccine, Rabies Vaccine for Human Use, Japanese Encephalitis Live Vaccine;
* You have accepted last immunization of Rabies Vaccine for Human Use after being bitten by an animal within 1 year;
* You have received the last vaccination of antitoxin or immune serum injection within 4 weeks, or got the last vaccination of hepatitis B human immunoglobulin within 1 year;
* You have been in a clinical trial within 6 months;
* You have clinical trial records within 3 months for the donation of WBC, plasma and platelet;
* You are evaluated by Investigator s as an unsuitable participant for this research.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Regardless of race and nationality, healthy subjects aged between 18 and 40 years old (including the tipping point), who have not previously donated blood.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-10-10 (Estimated); Primary Completion 2025-09-10 (Estimated); Study Completion 2025-09-10 (Estimated)

PRIMARY OUTCOMES:
Exploratory research and process development of immunocytotherapy-related products. | September10 2025
  Cultured cells under normal culture conditions or under the treatment of potential drug molecules, observe and record cell viability, proliferation, apoptosis, and functional expression.